CLINICAL TRIAL: NCT06589388
Title: ctDNA Monitoring to Predict the Efficacy of Total Neoadjuvant Therapy for Rectal Cancer
Brief Title: ctDNA Monitoring to Predict the Efficacy of TNT for Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Gene Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: GS_ZTR
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer; Rectal Cancer Stage II; Rectal Cancer Stage III
Keywords: liquid biopsy; circulating tumor DNA; Vietnam; total neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The 1st samples are collected from participants of Rectal cancer, phase II-III. They will be processed and analyzed to determine the detection rate of ctDNA in the blood samples before total neoadjuvant chemotherapy. The 2nd and 3rd samples collected from participants will be processed and analyzed to determine the change of ctDNA in the blood samples during and after total neoadjuvant therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study with three primary objectives:

Objective 1: Evaluate the detection rate and changes in circulating tumor DNA (ctDNA) levels in blood samples from colorectal cancer patients before, during, and after total neoadjuvant therapy (TNT).

Determine the detection rate and change of CtDNA in blood samples of cancer patients before, during, and after TNT then assess changes in ctDNA expression within the study population during treatment.

* Determine the ctDNA positivity rate before treatment.
* Determine the ctDNA positivity rate during TNT.
* Determine the ctDNA positivity rate after TNT and assess ctDNA level changes during treatment.

Objective 2: Investigate the relationship between ctDNA expression and MRI/CT scan imaging with the pathological complete response (pCR) to neoadjuvant therapy :

* Correlation between ctDNA detection and pCR/TRG/NAR score. Calculate the Positive Prediction Value - PPV, Negative Prediction Value - NPV of ctDNA,
* Correlation between MRI/CT scan imaging and pCR. Calculate the PPV and NPV of MRI/CT scan
* Combination of ctDNA detection and MRI/CT scan imaging to predict pCR. Calculate the PPV and NPV of the combined markers.

Objective 3: Evaluate the relationship between post-TNT ctDNA expression and disease-free survival in colorectal cancer patients.

DETAILED DESCRIPTION:
This is a prospective observational study conducted at the Medical Genetics Institute (MGI), in collaboration with 3 hospitals (175 Military Hospital, Nguyen Tri Phuong Hospital, and 108 Military Central Hospital). Participants must meet all inclusion criteria and no exclusion criteria (detailed in the eligibility section).

Sample Collection

* 10 mL of peripheral blood (Streck tubes) is collected for ctDNA analysis at 3 time points: pre-TNT (at diagnosis), middle of treatment (after chemoradiotherapy or after chemotherapy), and post-TNT (before surgery).
* 6-8 slides (6um thickness/slide) of FFPE biopsy tumor samples before treatment
* 6-8 slides (6um thickness/slide) of FFPE tumor samples collected after surgery. This sample is used to compare the mutational profiles with the corresponding biopsy samples.

Clinical results for collection

* Age, sex, medical history
* Number, size, and stage (TNM) of tumor
* MRI and/or CT scan images and reports at pre-treatment, mid-treatment, and end-treatment (before surgery)
* Histopathological evaluation of biopsy and surgery tissues, and conclusion of pathological response

  * TNM classification, pCR conclusion
  * TRG conclusion
* Disease-free survival follow-up for 2 years

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, both genders
* Patients are diagnosed with stage II-III rectal cancer and indicated for total neoadjuvant therapy
* Biopsy FFPE sample is available at the time of diagnosis
* Patients consented to participate in the study

Exclusion Criteria:

* Stage I rectal cancer, recurrent or metastatic cancer
* Other cancer metastasis to the rectum
* Patients are indicated for chemoradiation therapy only
* Have been or are being treated for cancer
* Patients do not agree to participate in the studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients aged 18 years and older, diagnosed with stage II-III rectal cancer, and indicated for total neoadjuvant chemotherapy. Participants must meet all inclusion criteria and no exclusion criteria. Recruitment will take place at 175 Military Hospital, Nguyen Tri Phuong Hospital, and 108 Military Center Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the detection rate and change of ctDNA in blood samples of rectal cancer patients during total neoadjuvant therapy | 12 months
  Determine the detection rate and change of CtDNA in blood samples of cancer patients before, during and after total neoadjuvant therapy and assess changes in ctDNA expression within the study population during treatment.
  * Determine the ctDNA positivity rate before treatment.
  * Determine the ctDNA positivity rate during total neoadjuvant therapy TNT.
  * Determine the ctDNA positivity rate after TNT and assess ctDNA level changes during treatment.
To investigate the relationship between ctDNA expression and MRI/CT scan imaging with pCR response in total neoadjuvant therapy (TNT) | 6 months
  * To investigate the prediction value of ctDNA to pathological complete response (pCR) in TNT: Calculate the percentage PPV, NPV of ctDNA to pCR
  * To investigate the prediction value of MRI/CT results to pCR in TNT: Calculate the percentage PPV, NPV of MRI/CT scan (RECIST 1.1) to pCR
  * To investigate the prediction value of MRI/CT results combined ctDNA results to pCR in TNT: Calculate the percentage PPV, NPV of MRI/CT combined ctDNA to pCR
Evaluate the relationship between post-TNT ctDNA expression and disease-free survival in colorectal cancer patients in 2 years | 24 months
  Create a Kaplan-Meier curve to estimate the disease-free survival of two years according to the after-treatment ctDNA status of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sinh D Nguyen, PhD, Principal Investigator — Medical Genetics Institude
Locations (1):
- Medical Genetics Institute, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data from this study may be requested for publication by journals. Sharing anonymized data with suitable studies will be decided by the sponsor, PIs, and the authority agency where the data was collected. No identifiable information will be shared with any other person/organization than authorized in the study.
Supporting Information: Study Protocol, ICF
Time Frame: Dec 2027
Access Criteria: GS_ZTR_ctDNA for Rectal Cancer

REFERENCES:
- [Background] Kim MJ, Lee DW, Kang HC, Park JW, Ryoo SB, Han SW, Kim KS, Chie EK, Oh JH, Jeong WK, Kim BH, Nam EM, Jeong SY. Total neoadjuvant therapy with short-course radiotherapy Versus long-course neoadjuvant chemoradiotherapy in Locally Advanced Rectal cancer, Korean trial (TV-LARK trial): study protocol of a multicentre randomized controlled trial. BMC Cancer. 2023 Aug 8;23(1):734. doi: 10.1186/s12885-023-11177-7. PMID 37553666
- [Background] Johnson GGRJ, Park J, Helewa RM, Goldenberg BA, Nashed M, Hyun E. Total neoadjuvant therapy for rectal cancer: a guide for surgeons. Can J Surg. 2023 Apr 21;66(2):E196-E201. doi: 10.1503/cjs.005822. Print 2023 Mar-Apr. PMID 37085291
- [Background] Lopez-Campos F, Martin-Martin M, Fornell-Perez R, Garcia-Perez JC, Die-Trill J, Fuentes-Mateos R, Lopez-Duran S, Dominguez-Rullan J, Ferreiro R, Riquelme-Oliveira A, Hervas-Moron A, Counago F. Watch and wait approach in rectal cancer: Current controversies and future directions. World J Gastroenterol. 2020 Aug 7;26(29):4218-4239. doi: 10.3748/wjg.v26.i29.4218. PMID 32848330
- [Background] Li LH, Chen ZF, Wang XF, Liu X, Jiang WZ, Zhuo SM, Jiang LW, Guan GX, Chen JX. Monitoring neoadjuvant therapy responses in rectal cancer using multimodal nonlinear optical microscopy. Oncotarget. 2017 Nov 3;8(63):107323-107333. doi: 10.18632/oncotarget.22366. eCollection 2017 Dec 5. PMID 29291032
- [Background] Feeney G, Sehgal R, Sheehan M, Hogan A, Regan M, Joyce M, Kerin M. Neoadjuvant radiotherapy for rectal cancer management. World J Gastroenterol. 2019 Sep 7;25(33):4850-4869. doi: 10.3748/wjg.v25.i33.4850. PMID 31543678
- [Background] Glynne-Jones R, Wyrwicz L, Tiret E, Brown G, Rodel C, Cervantes A, Arnold D; ESMO Guidelines Committee. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv22-iv40. doi: 10.1093/annonc/mdx224. No abstract available. PMID 28881920
- [Background] Hu H, Huang J, Lan P, Wang L, Huang M, Wang J, Deng Y. CEA clearance pattern as a predictor of tumor response to neoadjuvant treatment in rectal cancer: a post-hoc analysis of FOWARC trial. BMC Cancer. 2018 Nov 20;18(1):1145. doi: 10.1186/s12885-018-4997-y. PMID 30458734
- [Background] Yan YY, Guo QR, Wang FH, Adhikari R, Zhu ZY, Zhang HY, Zhou WM, Yu H, Li JQ, Zhang JY. Cell-Free DNA: Hope and Potential Application in Cancer. Front Cell Dev Biol. 2021 Feb 22;9:639233. doi: 10.3389/fcell.2021.639233. eCollection 2021. PMID 33693004
- [Background] McDuff SGR, Hardiman KM, Ulintz PJ, Parikh AR, Zheng H, Kim DW, Lennerz JK, Hazar-Rethinam M, Van Seventer EE, Fetter IJ, Nadres B, Eyler CE, Ryan DP, Weekes CD, Clark JW, Cusack JC, Goyal L, Zhu AX, Wo JY, Blaszkowsky LS, Allen J, Corcoran RB, Hong TS. Circulating Tumor DNA Predicts Pathologic and Clinical Outcomes Following Neoadjuvant Chemoradiation and Surgery for Patients With Locally Advanced Rectal Cancer. JCO Precis Oncol. 2021 Jan 12;5:PO.20.00220. doi: 10.1200/PO.20.00220. eCollection 2021. PMID 34250394
- [Background] Dizdarevic E, Hansen TF, Jakobsen A. The Prognostic Importance of ctDNA in Rectal Cancer: A Critical Reappraisal. Cancers (Basel). 2022 Apr 30;14(9):2252. doi: 10.3390/cancers14092252. PMID 35565381
- [Background] Nguyen Hoang VA, Nguyen ST, Nguyen TV, Pham TH, Doan PL, Nguyen Thi NT, Nguyen ML, Dinh TC, Pham DH, Nguyen NM, Nguyen DS, Nguyen DQ, Lu YT, Do TTT, Truong DK, Phan MD, Nguyen HN, Giang H, Tu LN. Genetic landscape and personalized tracking of tumor mutations in Vietnamese women with breast cancer. Mol Oncol. 2023 Apr;17(4):598-610. doi: 10.1002/1878-0261.13356. Epub 2023 Jan 15. PMID 36495126
- [Background] Nguyen HT, Nguyen TV, Nguyen Hoang VA, Tran DH, Le Trinh NA, Le MT, Nguyen Tran TA, Pham TH, Dinh TC, Nguyen TS, Nguyen The KC, Mai H, Chu MT, Pham DH, Nguyen XC, Ngo Ha TM, Nguyen DS, Nguyen DQ, Lu YT, Do Thi TT, Truong DK, Nguyen QT, Nguyen HN, Giang H, Tu LN. Tumor genomic profiling and personalized tracking of circulating tumor DNA in Vietnamese colorectal cancer patients. Front Oncol. 2022 Dec 12;12:1069296. doi: 10.3389/fonc.2022.1069296. eCollection 2022. PMID 36578946